CLINICAL TRIAL: NCT05936463
Title: The Effect of Clear Aligners and Metal Brackets on the Nutritional Status of Orthodontic Patients
Brief Title: Impact of Clear Aligners and Metal Brackets on Nutritional Status
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Marmara University (Other)
Responsible Party: Principal Investigator, Ferit Bayram, Assist. Prof., Marmara University
Other Study IDs: MUDHF_ORT_SBF_02
Record Dates: First submitted 2023-06-23; First posted 2023-07-07 (Actual); Last update posted 2023-07-10 (Actual); Status verified 2023-07

CONDITIONS: Malocclusion
Keywords: Tooth Crowding; Nutritional Status; Orthodontic Brackets; Clear Aligner Appliances
MeSH Terms: conditions — Malocclusion

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Orthodontics brackets
- Clear aligner appliances

SUMMARY:
This study aims to investigate the effect of clear aligners and traditional brackets on the nutritional status of orthodontic patients. With the increasing demand for more aesthetic and comfortable orthodontic appliances among adults, clear aligner treatment has gained popularity as an alternative to traditional fixed appliances. However, limited research has been conducted to evaluate the impact of clear aligners on dietary habits and nutrition. The study will include adult participants undergoing orthodontic treatment with either clear aligners or traditional brackets. Anthropometric measurements, dietary assessments, and oral health impact evaluations will be conducted to assess the nutritional status of the participants. The findings of this study will contribute to a better understanding of the influence of orthodontic appliances on nutrition and guide clinicians in providing comprehensive care to orthodontic patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult individuals (18 - 45 years old)
* Undergoing orthodontic treatment, without missing teeth in the mouth (excluding wisdom teeth)
* Having received orthodontic treatment for more than 6 months
* Citizens of the Republic of Turkey
* Proficient in reading and writing in the Turkish language
* Not under the influence of alcohol or drugs
* Able to understand and follow instructions for filling out the questionnaire
* Willing to participate in the study

Exclusion Criteria:

* Adult individuals (18 - 45 years old)
* Undergoing orthodontic treatment, without missing teeth in the mouth (excluding wisdom teeth)
* Having received orthodontic treatment for more than 6 months
* Citizens of the Republic of Turkey
* Proficient in reading and writing in the Turkish language
* Not under the influence of alcohol or drugs
* Able to understand and follow instructions for filling out the questionnaire
* Willing to participate in the study

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: The study population will consist of adult individuals aged 18-45 who are currently undergoing orthodontic treatment and do not have missing teeth (excluding wisdom teeth). They should have been receiving treatment for at least 6 months, be citizens of Turkey, proficient in Turkish language, and willing to participate. Exclusion criteria include age above 45, refusal to provide consent or answer all questions, specific dietary restrictions, eating disorders, pregnancy or breastfeeding, and cognitive impairment.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-04-01 (Estimated)

PRIMARY OUTCOMES:
Chewing Ability Assessment | Day 1
  Chewing ability will be evaluated using a questionnaire to assess both subjective and objective aspects. The questionnaire will consist of open-ended and closed-ended questions to determine individuals' chewing difficulties. Open-ended questions will focus on identifying specific foods that present challenges during chewing and the strategies employed to consume these foods. In subsequent follow-up interviews, closed-ended questions will be used to evaluate the ability to chew the previously listed foods, with response options such as "easy to chew," "experiencing some difficulty," and "experiencing great difficulty/cannot chew at all." If participants indicate experiencing slight or significant difficulty chewing at least two of the hard foods and four of the soft foods, it will be considered indicative of chewing difficulties. This assessment will provide valuable insights into the participants' chewing function and its impact on their dietary habits and oral health.
Oral Health Impact Profile-14 (OHIP-14) | Day 1
  The Oral Health Impact Profile-14 (OHIP-14) is a measurement tool developed to assess the impact of oral and dental health on individuals. It consists of 14 questions, and each question is rated on a scale of 0 to 4, with response options defined on a Likert scale as "0=never, 1=rarely, 2=sometimes, 3=often, and 4=always." The total score of OHIP-14 ranges from 0 to 56. A higher total score indicates increased severity of problems and decreased quality of life. In this study, OHIP-14 will be administered to participants to evaluate the impact of oral health on their daily functioning, well-being, and quality of life.

SECONDARY OUTCOMES:
Physical Activity Level | Day 1
  Physical activity levels of participants will be assessed using the International Physical Activity Questionnaire (IPAQ) short form. The IPAQ was developed with the support of the World Health Organization (WHO) and the Centers for Disease Control and Prevention (CDC), and its validity and reliability study was conducted in Turkey in 2010 by Sağlam et al. Individual Metabolic Equivalent Task (MET) scores will be calculated based on the IPAQ protocol to categorize participants into "low, moderate, and high activity levels." Total scores ranging from 0 to 600 will be classified as "low level," scores between 600 and 1500 or 3000 (depending on the number of days of moderate and vigorous physical activity per week) will be classified as "moderate level," and scores equal to or above 1500 or 3000 (depending on the number of days of moderate and vigorous physical activity per week) will be classified as "high level."
Height Measurement | Day 1
  The participants' height will be measured using standard procedures with the participants standing upright, heels together, head in an upright position, and looking straight ahead.
Body Composition | Day 1
  Body composition analysis will be performed with the Tanita DC-360 device that performs bioelectrical impedance analysis (BIA). The analysis report includes body weight (kg), body water mass (kg), body fat mass (kg) and body muscle mass (kg). This method is non-invasive and provides body composition data in less than 1 minute of measurement.
Waist Circumference | Day 1
  Waist circumference will be measured using a flexible tape measure placed horizontally around the smallest circumference between the lower rib and the iliac crest, parallel to the floor passing through the navel.

CONTACTS AND LOCATIONS:
Locations (1):
- Marmara University School of Dentistry, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided